CLINICAL TRIAL: NCT05255042
Title: Tissue Models for Liver Disease
Acronym: TIMOLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0814
Record Dates: First submitted 2022-01-06; First posted 2022-02-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Experiments include ex vivo liver segment perfusion and infection with bacteria or viruses. Biopsies of the perfused 24 liver segments are processed for in vitro tissue slice and macrophage cell culture. The resulting primary cell cultures and tissue slices will be stored frozen for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial Participants: Overall Description of Trial Participants: The liver organ samples included in this project will be from patients undergoing elective surgery for a lesion in the liver in the HPB Unit of the Leicester General Hospital. No change in the surgical procedure or recruiting results from this study and the use of the samples.
  Inclusion Criteria: The samples included in this project will be from patients undergoing elective liver surgery in the HPB Unit of the Leicester General Hospital. The criteria for inclusion of liver segment samples from radical surgery are adult age and presence of hepatic tissue in the discarded material after hepato-pancreato-biliary surgery.
  Exclusion Criteria: The main exclusion criterion is acute invasive infection, but these patients are automatically excluded from major surgery. Vulnerable groups will not be recruited.
  Interventions: Other: organ and tissue sample collection only

INTERVENTIONS:
Other: organ and tissue sample collection only — Collection of liver segments removed by radical surgery of hepatic lobes, but not submitted to pathology

SUMMARY:
The human immune response to bacterial and viral local and systemic infection are fairly well understood, but we lack details on the earliest phases. Better knowledge of these events would be important for the prevention and treatment of severe bacterial or viral disease. From models of infection, we have data showing that bacteria replicate in a specific type of cells in the liver from where the bacteria then seed to the blood to cause blood stream infection. In order to gain more relevant data for humans, we have developed a spleen and liver perfusion model using pig organs. This model confirms our previous work and most importantly will now allow us to study these events in human organs.

Primary Objectives: The primary objective of the study is to identify therapies acting on the initial events during invasive bacterial and viral infection.

Secondary Objectives: The secondary objective of this study is to provide novel in vitro and ex vivo models of human liver macrophages to study the impact of therapies for invasive infection.

The Primary Endpoint of the study is to increase the resistance of liver macrophages to infection at least tenfold after treatment.

The Primary Outcome Measure of the study is the reduction of bacterial or viral load at pre-determined time-points.

DETAILED DESCRIPTION:
This is a preclinical research project and no patient intervention is planned. The project makes use of anonymised human tissue samples discarded during radical surgery. The liver segment samples included in this project will be from patients undergoing elective surgery for a lesion in the liver in the HPB Unit of the Leicester General Hospital. The sample size of 96 patiens (46 liver segments) has been determined by power calculations and is in line with the number of livers actually removed by elective liver surgery over the past years. No change in the surgical procedure or recruiting results from this study and the use of the samples. All the experimental work carried out on the liver samples will have no effect on the patient.

Experiments include ex vivo organ segment perfusion and infection with bacteria or viruses. Biopsies of the perfused 46 liver segments are processed for in vitro tissue slice and macrophage cell culture. The resulting primary cell cultures and tissue slices will be stored frozen for future research. All in vitro studies on the 46 liver segments, and the tissues and cells derived from them, will evaluate the effect of therapeutic interventions (antibodies, receptor antagonists, antibiotics and other molecules) on the capacity of liver cells to clear invasive bacteria or viruses. The experiments will be carried out each time a liver sample will be available.

The detailed technical description of the experimental strategy including the strategy for storage and discarding of the human tissue will be as follows:

1. Liver segment ex vivo perfusion: This work is done to stabilise the organ, infect the organ and then to derive from it tissue slices and cells for primary cell culture. We have successfully set up a normo-thermic ex vivo porcine liver perfusion model. This expertise allowed us to define the parameters for organ collection, transport and perfusion of porcine livers for up to twenty-four hours and importantly develop and infection model. Infection showed conservation of capacity to remove bacteria from blood and good filtering capacity and, essential for this application, that also in the whole organ model specific subsets of macrophages are permissive to bacterial intracellular replication. In this experimental series we propose to perfuse explanted human liver segments. In contrast to pigs, we will use for perfusion of the human organ synthetic medium in order to neutralise or minimise acquired immunity. Histology, confocal microscopy, FACS analysis and bacterial and viral enumeration will be the main methodologies to analyse the perfused organ. The aim of this part of the work is to demonstrate that at the organ level bacteria and viruses are able to replicate in liver tissue macrophages pinpointing attention of anti-infective treatments to the prevention of these early steps potentially preventing invasive bacterial and viral disease. Samples from the 46 perfused organ segments will be the source of tissue slice cultures and primary cell cultures.
2. Primary cell cultures: From the 46 human liver segments we will derive samples for primary culture of human tissue macrophages and other immune cells. Using the methodology in use for cells from mice and pigs, we will set up primary cultures of human hepatic immune cells and in particular macrophages. Immune cells including macrophages and neutrophils will be purified by different methodologies including by percoll gradient centrifugation, FACS and magnetic separation and cultured for up to seven days. Cultures will be tested for multiple parameters including cytokines, surface markers, anybody production and gene expression. To test interaction with bacteria or viruses, the cultured cells will be infected with a panel of bacterial and viral pathogens. Upon other methodology, confocal microscopy, FACS and RNAseq will be used monitor behaviour of bacterial and viral pathogens and host cells. Interventions with cytokines, chemokines, drugs, antibiotics and other compounds will be carried out to test tractability of the system. No genotyping of the organ will be performed. With the aim in mind to identify targets for intervention, the cell culture models are intended to provide detailed quantifiable parameters of the interaction of bacteria or viruses and immune cells in particular tissue macrophages in a controlled in vitro culture system. This is intended to allow the design of medium-throughput assays to test strategies modifying initiation of invasive disease. Cells will be stored in liquid nitrogen for further research.
3. Organotypic slice cultures: From the 46 human liver segments we will derive, in addition to cells, also tissue samples for organotypic slice cultures. With the methodology well set up for brain slices and described for liver, we will culture organotypic human liver slice cultures. These organ slices are superior to cell cultures, as they maintain the multicellular spatial microarchitecture of the organ, which is particularly important when analysing tissue macrophages. As for brain slice cultures, we will infect the slices with bacterial or viral pathogens and monitor their migration within the tissue, the infection of cells and the reaction of the single host cells. The use of tissue slice culture should allow to specifically study the targeting and replication-permissive nature of specific subsets of immune cells including macrophages. A goal of the objective is to allow for detailed development of infectious foci in the liver including time laps confocal microscopy of infected liver slices. Testing in this model cytokines and other host derived molecules are expected to show the potential of interventions targeting specific subsets of immune cells including macrophages. Tissue slices will be stored in liquid nitrogen for further research.

ELIGIBILITY:
Inclusion Criteria:

* The samples included in this project will be from patients undergoing elective surgery in the HPB Unit of the Leicester General Hospital.
* Liver segment samples from radical surgery are adult age (18-80 years)
* Presence of liver segment tissue in the discarded material after hepatopancreato-biliary surgery.

Exclusion Criteria:

* The main exclusion criterion is acute invasive l infection, but these patients are automatically excluded from major surgery.
* Samples from patients treated with antibiotics prior to explant or surgery will not be excluded, but samples will have to be tested for residual antibiotic activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The liver segment samples included in this project will be from patients undergoing elective surgery for a lesion in the liver in the HPB Unit of the Leicester General Hospital. No change in the surgical procedure or recruiting results from this study and the use of the samples.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of the load and replication of infectious agents by host directed interventions | 3.5 Years
  Reduction of the number of infectious agents per gram of tissue by therapies acting on the initial events during invasive infection.

SECONDARY OUTCOMES:
Protocol for seven-day survival of tissue slices and primary macrophage cell cultures | 3.5 Years
  Protocol for seven-day survival of tissue slices and primary macrophage cell cultures to study in vitro therapies for invasive infection

CONTACTS AND LOCATIONS:
Overall Officials: Marco R Oggioni, MD, Principal Investigator — University of Leicester
Locations (1):
- UHL NHS Trust - Leicester General Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wanford JJ, Hames RG, Carreno D, Jasiunaite Z, Chung WY, Arena F, Di Pilato V, Straatman K, West K, Farzand R, Pizza M, Martinez-Pomares L, Andrew PW, Moxon ER, Dennison AR, Rossolini GM, Oggioni MR. Interaction of Klebsiella pneumoniae with tissue macrophages in a mouse infection model and ex-vivo pig organ perfusions: an exploratory investigation. Lancet Microbe. 2021 Dec;2(12):e695-e703. doi: 10.1016/S2666-5247(21)00195-6. PMID 34901898
- [Background] Carreno D, Wanford JJ, Jasiunaite Z, Hames RG, Chung WY, Dennison AR, Straatman K, Martinez-Pomares L, Pareek M, Orihuela CJ, Restrepo MI, Lim WS, Andrew PW, Moxon ER, Oggioni MR. Splenic macrophages as the source of bacteraemia during pneumococcal pneumonia. EBioMedicine. 2021 Oct;72:103601. doi: 10.1016/j.ebiom.2021.103601. Epub 2021 Oct 4. PMID 34619637